CLINICAL TRIAL: NCT02426697
Title: Phase 3 Study Evaluating Fentanyl Transmucosal in the Prevention of Pain Induced by Mobilization During Radiotherapy in Patients With Bone Metastasis
Brief Title: Pain Management With Pecfent in the Prevention of Pain Induced by Position in Radiotherapy
Acronym: PARABONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHB14.03
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Bone Metastasis
Keywords: bone metastasis, radiotherapy, pain, prevention
MeSH Terms: conditions — Pain | interventions — Fentanyl; Administration, Mucosal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pecfent (Experimental): Patients will receive 100 µg of transmucosal Pecfent before radiotherapy session (or 200 µg in patients with a stable opioid background pain treatment)
  Interventions: Drug: fentanyl transmucosal
- Placebo (Placebo Comparator): Patients will receive 100 µg of transmucosal placebo before radiotherapy session or 200 µg in patients with a stable opioid background pain treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fentanyl transmucosal — Participation to the trial will be proposed to the patient by the investigator in charge of the analgesic irradiation during preliminary scanner session. When starting the radiotherapy session, investigator will collect the signed inform consent form, deliver the treatment, will collect pain intensity value using VAS (before and after the radiotherapy session).
  Other Names: Pecfent
  Arms: Pecfent
Drug: Placebo — Participation to the trial will be proposed to the patient by the investigator in charge of the analgesic irradiation during preliminary scanner session. When starting the radiotherapy session, investigator will collect the signed inform consent form, deliver the treatment, will collect pain intensity value using VAS (before and after the radiotherapy session).
  Other Names: Placebo in transmucosal use
  Arms: Placebo

SUMMARY:
The clinical trial is a stage 3 study to determine the role of fentanyl transmucosal in the prevention of pain induced by mobilization in patients receiving a bone metastasis radiation for bone metastasis irradiations

DETAILED DESCRIPTION:
Participation to the trial will be proposed to the patient by the investigator in charge of the analgesic irradiation during the preliminary scanner session that will be held before radiotherapy session(s). Patients with a VAS≤ 3 will be excluded.

PecFent and Placebo will be delivered by Archimedes Pharma When starting the radiotherapy session(s) (2 days after the preliminary scanner session), the medic will collect the patient signed informed consent, will deliver the treatment 1 dose of fentanyl transmucosal (Pecfent® ) 100µg in naive patients or 1 dose of Pecfent® 200µg in patient with a stable opioid background pain treatment or placebo) and will collect pain intensity value with a patient VAS collected before and at the end of the radiotherapy session. Finally patient & radiotherapists global satisfaction will be collected An assessment a week the end of the radiotherapy session will be assessed by investigator consisting in a Patient global satisfaction

Study follow up:

Patients will receive a phone call a week after the radiotherapy session to collect patient global satisfaction score related with the global management of the radiotherapy session

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* More than 18 years old
* Proven histological cancer with bone metastasis
* SignedInform consent form
* Patient with pain assed as VAS Superior to 3 when positioning the patient in the preliminary scanner session

Exclusion Criteria:

* VAS>3 before radiotherapy treatment (establishment of an appropriate analgesic treatment) (session
* Any SAO treatment on going
* Pregnant or lactating woman
* Hypersensitivity or safety issues to any opioïd treatment
* Poor nasal mucosa (defined on clinical doctor assessment)
* Severe obstructive lung conditions or respiratory depression
* Renal insufficiency with creatinine clearance inferior to 45 ml/min
* Hepatic insufficiency
* Patient misunderstanding of the content and objective of the trial
* Patient under supervision or guardianship
* SAO intake 4 hours before the radiotherapy session
* Patient participating to any other pain management trial
* Morphine pump usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Drug efficacy | 30 minutes
  Pain Intensity Difference (PID) with the VAS considering the higher Pain Intensity (PI) score notified by the patient during the scanner and radiotherapy session

SECONDARY OUTCOMES:
Patient global satisfaction | one week
  - Patient Global Satisfaction Score [0 (not satisfied) to 5 (very satisfied) one week after the radiotherapy session. Patients will receive a phone call a week after the radiotherapy session to collect patient global satisfaction score related with the global management of the radiotherapy session
Adverse event of Pecfent | one week
  Percentage of patient with side effects due to Pecfent
Rescue medication | 30 minutes
  Percentage of patients needing rescue medication during radiotherapy session
Radiotherapy session duration | one hour
  Duration of the session between the patient is discharged from the cabin until his return in the cabin

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Thureau, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France